CLINICAL TRIAL: NCT04447833
Title: Mesenchymal Stromal Cell Therapy For The Treatment Of Acute Respiratory Distress Syndrome Validation of Mechanistic Pathways and Clinical Efficacy
Brief Title: Mesenchymal Stromal Cell Therapy For The Treatment Of Acute Respiratory Distress Syndrome
Acronym: ARDS-MSC-205
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02238
Record Dates: First submitted 2020-06-20; First posted 2020-06-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: ARDS, Human; COVID
Keywords: Mesenchymal Stromal Stem Cells
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: This is an open label, dose escalating safety study of the advanced therapy investigational medicinal product (ATIMP) KI-MSC-PL-205, where patients diagnosed with SARS-CoV-2-induced severe acute respiratory distress syndrome (ARDS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stromal Stem Cell Treatment (Experimental): Infusion of allogeneic bone marrow derived mesenchymal stromal stem cells (MSC). First three patients receive a singe dose of 1x10^6 MSC/kg dose, next six patients receive a single dose of 2x10^6 MSC/kg.
  Interventions: Drug: Mesenchymal Stromal Stem Cells - KI-MSC-PL-205

INTERVENTIONS:
Drug: Mesenchymal Stromal Stem Cells - KI-MSC-PL-205 — Allogeneic bone marrow derived mesenchymal stromal stem cells (MSCs).
  Other Names: Allogeneic Bone Marrow Derived Mesenchymal Stem Cells

SUMMARY:
This is an open label, dose escalating safety study of the advanced therapy investigational medicinal product (ATIMP) KI-MSC-PL-205, where patients diagnosed with SARS-CoV-2-induced severe acute respiratory distress syndrome (ARDS), according to the Berlin Definition, and who are on respirator/ventilator (used synonymously in this protocol) support due to respiratory insufficiency with or without concomitant circulatory problems, will be included and treated with a single dose of KI-MSC-PL-205.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to performing study procedures (and have given written consent)
* Coronavirus (SARS-CoV-2) infection confirmed by polymerase chain reaction (PCR) test at screening
* Male or female patient aged 18 to 65 years old
* Patient must fulfil the Berlin Definition of severe ARDS within 3 weeks to 48 hours prior to enrolment (Will be assessed once the patient has been admitted to the ICU)
* Patient is on respirator support within 3 weeks to 48 hours prior to enrolment (Will be assessed once the patient has been admitted to the ICU)
* Pregnancy test in blood confirming negative results before enrolment (for women ≤55 years old)

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study
* Patients with history of treated blood and/or solid organ malignancy with recurrence within five years prior to dosing of the ATIMP are to be excluded. Patients with history of cervix cancer and non-melanoma skin cancer with recurrence within two years prior to dosing of the ATIMP are to be excluded
* Pregnant or breast feeding female
* Patient with a history of anti-coagulation therapy for other indications that short-term prophylaxis after surgery
* Patients with a history and/ or on-going treatment for entity associated with bleeding disorder or potential risk for bleeding (e.g. inflammatory bowel disease, gastro-esophagitis with or without ulcers, haemophilia and other bleeding disorders, inflammatory musculo-skeletal disease with potential bleeding complications)
* Patients with a history during the latest five years and/or on-going treatment for systemic infection (e.g. Septicaemia due to in vivo foreign body (e.g. stents, catheters, heart valve), tuberculosis, malaria, other opportunistic and parasite infections)
* Prisoner
* Any other irreversible disease or condition for which six-month mortality is estimated to be greater than 50%
* Moderate to severe liver failure (Child-Pugh Score >12)
* Reduced renal function with a creatinine clearance (Cockcroft-Gault Equation) < 45 mL/min/1.73m2
* Severe chronic respiratory disease with a PaCO2 >50 mmHg or the use of home oxygen
* Major trauma in the prior 5 days
* Lung transplant patient
* Patients on ECMO-support
* Patients with a previous history of severe burns
* Documented deep venous thrombosis or pulmonary embolism within past three months
* Known hypersensitivity to DMSO
* Investigator considers the patient unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of pre-specified treatment related adverse events of interest (TRAEIs). | From drug administration to day 10 post-infusion
  The incidence of pre-specified treatment related adverse events of interest (TRAEIs) occurring during the 10 days interval beginning with the start of the ATIMP infusion:
  * New ventricular tachycardia, ventricular fibrillation or asystole within 10 days after infusion
  * New cardiac arrhythmia requiring cardioversion within 10 days after infusion
  * Clinical scenario consistent with transfusion incompatibility or transfusion-related infection within 10 days after infusion
  * Thromboembolic events (e.g. Pulmonary embolism) within 10 days after infusion
  * Cardiac arrest or death within 10 days after infusion

SECONDARY OUTCOMES:
Safety; All-cause mortality | 60 days post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  All-cause mortality at 60 days and then annually
Changes in Leucocytes | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in the leucocyte Count (number/L)
Changes in Trombocytes | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in the trombocyte Count (number/L)
Changes in plasma concentration of C-reactive protein (CRP) | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in the plasma concentration of CRP (mg/L)
Changes in plasma concentration of Prothrombin complex (PK) | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in the plasma concentration of PK (INR)
Changes in plasma concentration of Creatinine | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in the plasma concentration of creatinine (μmol/L)
Changes in plasma concentration of Aspartate amino transferase (ASAT) | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in the plasma concentration of ASAT (μkat/L)
Changes in plasma concentration of Alanine amino transferase (ALAT) | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in the plasma concentration of ALAT (μkat/L)
Changes in plasma concentration of N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in the plasma concentration of NT-proBNP (ng/L)
Changes in Blood pressure | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in blood pressure (mmHg)
Changes in Body temperature | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in body temperature (°C)
Efficacy; Changes in pulmonary compliance | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in pulmonary compliance (dynamic and static) until day 10 post-infusion
Efficacy; Changes in driving pressure (Plateau pressure- PEEP) | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in driving pressure (Plateau pressure- PEEP) until day 10 post-infusion
Efficacy; Changes in oxygenation (PaO2/FiO2) | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion
  Changes from baseline (Day 1; prior to administration of ATIMP) in oxygenation (PaO2/FiO2) until day 10 post-infusion
Efficacy; Duration of ventilator support | Baseline (pre-infusion),day 1, 2, 3, 4, 7, 10 and 60 post-infusion
  Number of days with ventilator support
Efficacy; Pulmonary bilateral infiltrates | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes in amount of pulmonary bilateral infiltrates assessed by pulmonary X-ray from baseline (Day 1; prior to administration of ATIMP) until day 60
Efficacy; Sequential Organ Failure Assessment (SOFA) score | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, end of ICU
  Changes in Sequential Organ Failure Assessment (SOFA) score from baseline (Day 1; prior to administration of ATIMP) and during the ICU-period
Efficacy; Hospital stay | Day 60 post-infusion
  Duration of ICU stay and hospital stay (number of days; whole hospital period + calculated from Day 1)
Lung function | Day 60 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Recovery of lung function assessed by Spirometry (FEV1, Vital Capacity) at day 60 and then annually
Lung fibrosis | Baseline (pre-infusion), day 1, 3, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  To assess development of lung fibrosis using the HRCT Fibrosis Score using Computed tomography (CT) at baseline and on day 1, 3, 7, 10, end of ICU-residence, end of hospital stay, day 60, 6 month and 12 month and end of study (if possible during the infectious stage depending on hospital safety regimen during the pandemic).
Six minutes walk test | 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Assessment of the patient's physical capacity by 6-Minute-Walk-Test (6MWT), starting at 6 months post Day 1 and then annually
Changes in Quality of life | 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Changes in Quality of Life by assessing the Short Form Health Survey (SF-36) score (starting at 6 months post Day 1 and then annually; patient reported outcome)
Blood biomarkers | Baseline (pre-infusion), day 1, 2, 3, 4, 7 and 10 post-infusion, 6 months, 1, 2, 3, 4 and 5 years post-infusion
  Change in blood biomarkers related to the proposed mechanisms of action of KI-MSC-PL-205 in ARDS
Sensitisation test | Baseline (pre-infusion), day 60 post-infusion
  Sensitisation tests (test for donor-specific antibodies) against KI-MSC-PL-205 donor

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Simonsson, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden